CLINICAL TRIAL: NCT02285686
Title: Prognostic Value of Elevated Troponins in Critical Illness Study: A Pilot Study
Acronym: PRO-TROPICS
Status: Completed | Type: Observational
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: 14-674; 14348 (Other Grant/Funding Number: Hamilton Health Sciences - New Investigator Fund)
Record Dates: First submitted 2014-11-05; First posted 2014-11-07 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Troponin; Critical Care; Myocardial Infarction
Keywords: troponin; biomarkers; myocardial infarction; critical illness
MeSH Terms: conditions — Myocardial Infarction; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 2 cryovials
Oversight: Data Monitoring Committee: No

SUMMARY:
Troponins are sensitive and specific markers of cardiac injury. Critically ill patients frequently have elevated troponins. In this population, distinguishing patients with elevated troponins from those with myocardial infarction is difficult. However, troponin elevations on their own seem to be associated with an increased risk of death. The optimal treatment of patients with type 2 myocardial infarction or non ischemia related troponin elevations during critical illness is unclear. There are no trials in the ICU setting to guide management.

This study is a 1-month pilot cohort study of troponin screening in 4 Ontario intensive care units. The objective of this pilot study is to evaluate the ability to perform a larger study, which will determine the prevalence, incidence and risk factors for elevated troponin values, how patients with elevated troponin values are treated as a baseline, and the incidence of myocardial infarction in critically ill patients. Knowing the prognostic impact of these conditions and understanding current management will thereafter guide researchers and clinicians on the importance of carefully evaluating potential risk-modifying therapies.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients admitted to the participating ICUs of study sites during the study enrollment period will be eligible.

Exclusion Criteria:

* Patients who are admitted and die or are discharged within 12 hours
* Patients re-admitted to ICU during the index ICU enrolment month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients
Sampling Method: Non-Probability Sample
Enrollment: 251 (Actual)
Dates: Start 2014-11; Primary Completion 2015-03-15 (Actual); Study Completion 2015-03-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | 1 month
  Feasibility outcome
Data collection time per patient | 3 months
  Feasibility outcome
rate of successful deferred informed consent definition | 1 month
  Feasibility outcome

SECONDARY OUTCOMES:
All-cause in-hospital mortality | 3 months
Troponin elevations | 3 months
Myocardial infarction | 3 months